CLINICAL TRIAL: NCT00002032
Title: Rifabutin Therapy for the Prevention of Mycobacterium Avium Complex (MAC) Bacteremia in AIDS Patients With CD4 Counts = or < 200: A Double-Blind, Placebo-Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 048A; 087023-999
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-01

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Antitubercular Agents
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Rifabutin

INTERVENTIONS:
Drug: Rifabutin

SUMMARY:
The primary objectives of this trial are: To compare the safety of oral rifabutin versus placebo in the treatment of Mycobacterium avium complex (MAC) bacteremia in AIDS patients with CD4 counts less than or equal to 200 cells/mm3. To investigate the incidence of MAC in these patients. A secondary objective is to compare clinical response, quality of life (Karnofsky), and survival between these two groups.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Diagnosis of AIDS with a case defining infection other than Mycobacterium avium complex (MAC).
* Written informed consent.
* Females of childbearing potential must also sign a special informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Known hypersensitivity to rifabutin, rifampin, other rifamycins, zidovudine or didanosine (ddI).
* Previous or current infection due to Mycobacterium avium complex (MAC) disease as evaluated by two successive blood cultures and two successive stool cultures taken within 14 days prior to study initiation.

Concurrent Medication:

Excluded:

* Antiretroviral agents other than zidovudine (AZT).
* Didanosine (ddI).
* Antimycobacterial therapy.
* Rifampin.
* Isoniazid.
* Clofazimine.
* Ethambutol.
* Cycloserine.
* Ethionamide.
* Amikacin.
* Ciprofloxacin.
* Streptomycin.
* Other investigational drugs.
* If antimicrobial therapy is required to treat bacterial infections (= or < 14 days), Adria Laboratories must be contacted prior to initiation of therapy.

Patients with the following are excluded:

* Known hypersensitivity to rifabutin, rifampin, other rifamycins, zidovudine (AZT), or didanosine (ddI).
* Previous or current Mycobacterium avium complex (MAC) infection.
* Perceived patient unreliability or unavailability for frequent monitoring.

Prior Medication:

Excluded within 4 weeks of study entry:

* Antiretroviral agents other than zidovudine (AZT) or didanosine (ddI).
* Antimycobacterial therapy.
* Rifampin.
* Isoniazid.
* Clofazimine.
* Ethambutol.
* Cycloserine.
* Ethionamide.
* Amikacin.
* Ciprofloxacin.

Required:

* Zidovudine (AZT).
* Antipneumocystis prophylactic therapy.

Required for at least 4 weeks prior to study entry:

* Zidovudine (AZT) or didanosine (ddI).
* Antipneumocystis prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Ctr for Special Immunology, Irvine, California
  - Olive View Med Ctr, Sylmar, California
  - Denver Public Health Dept, Denver, Colorado
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Ctr for Special Immunology, Fort Lauderdale, Florida
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Mem Hosp Hollywood, Hollywood, Florida
  - VP Med Services / HHCS Research Institute Inc, Orlando, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Grady Memorial Hosp / Hughs Spalding Med Ctr, Atlanta, Georgia
  - Dr Winkler Weinberg, Roswell, Georgia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - CRI of New England, Brookline, Massachusetts
  - Univ of Missouri at Kansas City School of Medicine, Kansas City, Missouri
  - Research Med Ctr, Kansas City, Missouri
  - Brooklyn Veterans Administration, Brooklyn, New York
  - Maimonides Med Ctr, Brooklyn, New York
  - Nassau County Med Ctr, East Meadow, New York
  - Long Island Jewish Med Ctr, New Hyde Park, New York
  - Community Research Initiative, New York, New York
  - Chelsea Village Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Med Ctr, Columbus, Ohio
  - Central Texas Med Foundation, Austin, Texas
  - Nelson Tebedo Community Clinic, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Texas Tech Health Sciences Ctr, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Univ TX San Antonio Health Science Ctr, San Antonio, Texas
  - Scott and White Hosp, Temple, Texas
  - Dr Scott Lea, Waco, Texas

REFERENCES:
- [Background] Dautzenberg B, Castellani P, Pellegrin JL, Vittecoq D, Truffot-Pernot C, Pirotta N, Sassella D. Early bactericidal activity of rifabutin versus that of placebo in treatment of disseminated Mycobacterium avium complex bacteremia in AIDS patients. Antimicrob Agents Chemother. 1996 Jul;40(7):1722-5. doi: 10.1128/AAC.40.7.1722. PMID 8807071
- [Background] Moore RD, Chaisson RE. Survival analysis of two controlled trials of rifabutin prophylaxis against Mycobacterium avium complex in AIDS. AIDS. 1995 Dec;9(12):1337-42. doi: 10.1097/00002030-199512000-00006. PMID 8605053